CLINICAL TRIAL: NCT02860572
Title: Non-interventional Follow-up Versus Fluid Bolus in RESPONSE to Oliguria in the Optimization Phase of Fluid Therapy in the Critically Ill (the RESPONSE Trial)
Brief Title: Non-interventional Follow-up Versus Fluid Bolus in RESPONSE to Oliguria in the Critically Ill
Acronym: RESPONSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helsinki University Central Hospital (Other)
Collaborators: Central Finland Central Hospital (Unknown)
Responsible Party: Principal Investigator, Suvi Vaara, MD, PhD, Helsinki University Central Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 200/13/03/02/16
Record Dates: First submitted 2016-08-01; First posted 2016-08-09 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Critically Ill; Acute Kidney Injury; Sepsis; Oliguria
Keywords: fluid therapy; oliguria; endothelial injury
MeSH Terms: conditions — Critical Illness; Acute Kidney Injury; Sepsis; Oliguria | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- follow-up without intervention (Experimental): No intervention to increase the urine output within 2 hours will be done.
  Interventions: Other: follow-up without intervention
- Standard group - fluid bolus (Active Comparator): Patient will receive 500mL of balanced crystalloid intravenously over 30 minutes.
  Interventions: Other: fluid bolus

INTERVENTIONS:
Other: follow-up without intervention
  Arms: follow-up without intervention
Other: fluid bolus
  Arms: Standard group - fluid bolus

SUMMARY:
Background: After hypotension, oliguria (urine output less than 0.5 mL/kg/h) was the most common trigger to administer fluid bolus in a multinational practice survey in intensive care. The effect of fluid bolus on cardiovascular variables can be very short-lived among patients in shock suggesting that fluid boluses in the optimization phase are unlikely to improve patient-centered outcomes. Moreover, a growing body of evidence suggests a poor renal response to fluid bolus.

Objective: To investigate, whether fluid bolus - as a standard of care - improves urine output in oliguric patients compared to a non-interventional follow-up approach without fluid bolus.

Design: Investigator-initiated, open, randomized, controlled study

Interventions:

1. Intervention group - follow-up without intervention
2. Control group - fluid bolus (500mL of balanced crystalloid over 30 minutes)

Randomization: 1:1 stratified according to the site, presence of acute kidney injury, and sepsis

Trial size: 130 patients randomized in 2 ICUs

DETAILED DESCRIPTION:
Study hypothesis:

The investigators hypothesize that fluid bolus given due to oliguria does not improve urine output in a majority of patients, especially among those with acute kidney injury. Another study hypothesis is that patients receiving fluid bolus will have higher levels of endothelial damage biomarkers.

Intervention description:

Intervention group -follow-up without intervention; No intervention to increase the urine output within 2 hours will be done.

Standard group - Fluid bolus group: Patient will receive 500mL of balanced crystalloid intravenously over 30 minutes.

In both groups, if severe hemodynamic instability occurs, a rescue bolus of 500mL over 30 minutes may be given according to the decision of the treating clinician.

In both groups, all other ongoing infusions (nutrition and on-going clear fluids) will be held constant during the 2-hour period. Vasoactive medications, sedation, short-acting insulin, and other medications can be modified according the clinical need. No diuretics during the 2-hour study period are allowed. After two hours from randomization, treating clinician can modify the fluid and drug therapy according to the clinical needs of the patient. All administered fluids will be recorded 6 h from randomization.

Except for the study intervention period of 2 hours, no attempt to control fluid therapy will be done. During the study period, all other aspects of critical care will follow the ICU's standard operating procedures and clinician's prescription.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18
* Emergency admission to an ICU
* Mean arterial pressure (MAP) >65 mmHg (with vasopressors if needed) and initial fluid resuscitation for shock/hypovolemia has been given
* Oliguria (urine output less than 0.5mL/kg/h) for at least 2 consecutive hours

Exclusion Criteria:

* Marked fluctuations in hemodynamics within last 2 hours (cardiac arrhythmias, increase in norepinephrine need over 0.2ug/kg/min, need for initiation of inotrope/inodilator)
* Administration of furosemide within last 6 hours
* Chronic kidney disease (estimated pre-critical illness GFR < 60ml/min/1.73m2)
* Renal replacement therapy
* Among patients with acute kidney injury, urgent indications for commencing renal replacement therapy
* Fluid overload (cumulative fluid accumulation exceeds 10% of baseline body weight)
* Pulmonary edema (bilateral infiltrates in chest x-ray)
* Active bleeding (need for transfusion, platelets, or fresh frozen plasma)
* Suspected or known intra-abdominal hypertension (IAP >16mmHg)
* Pregnant or lactating
* Expected survival less than 24h
* Obtaining informed consent is not possible/consent is denied

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2017-01-10 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2020-12-10 (Actual)

PRIMARY OUTCOMES:
Change in individual mean cumulative urine output (mL/kg/h) | 2 hours after randomization compared to urine output 2 hours preceding randomization
  Doubling of the urine output is defined as clinically meaningful response

SECONDARY OUTCOMES:
The difference between groups in the change in individual urine output | 2 hours after randomization compared to urine output 2 hours preceding randomization
Duration of consecutive oliguria (urine output <0.5 mL/kg) | during ICU stay, i.e. as long as urine output stays below 0.5 mL/kg/h while the patient is in the ICU (an average of 5 to 7 days) or until renal replacement therapy is commenced
Cumulative fluid balance | six hours from randomization

OTHER OUTCOMES:
Number of patients receiving rescue boluses and the number of rescue boluses | study intervention period (i.e. 2 hours)
Highest stage of acute kidney injury | within 24 hours, 48 hours and during ICU stay (an average of 5 to 7 days or up to 30 days if patient is still in ICU)
Number of patients with one or several protocol violation(s) and number of those per patient | study intervention period (i.e. 2 hours)
Number of patients with adverse events | from randomization to next morning
Number of patients receiving renal replacement therapy | during ICU stay(an average of 5 to 7 days or up to 30 days if patient is still in ICU)
change in mean arterial pressure | from randomization to 2 hours post-randomization
change in heart rate | from randomization to 2 hours post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Suvi Vaara, MD, PhD, Principal Investigator — Helsinki University Central Hospital
Locations (2):
- Finland (2):
  - Helsinki University Hospital, Meilahti, Helsinki, Uusimaa
  - Central Finland Central Hospital, Jyväskylä

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Serlo M, Inkinen N, Lakkisto P, Valkonen M, Pulkkinen A, Selander T, Pettila V, Vaara ST. Fluid bolus increases plasma hyaluronan concentration compared to follow-up strategy without a bolus in oliguric intensive care unit patients. Sci Rep. 2024 Sep 6;14(1):20808. doi: 10.1038/s41598-024-71670-2. PMID 39242877
- [Derived] Inkinen N, Pettila V, Valkonen M, Serlo M, Backlund M, Hastbacka J, Pulkkinen A, Selander T, Vaara ST. Non-interventional follow-up versus fluid bolus in RESPONSE to oliguria in hemodynamically stable critically ill patients: a randomized controlled pilot trial. Crit Care. 2022 Dec 22;26(1):401. doi: 10.1186/s13054-022-04283-8. PMID 36550559
- [Derived] Inkinen N, Selander T, Pettila V, Valkonen M, Backlund M, Wennervirta J, Pulkkinen A, Hastbacka J, Vaara ST. Noninterventional follow-up vs fluid bolus in RESPONSE to oliguria-The RESPONSE trial protocol and statistical analysis plan. Acta Anaesthesiol Scand. 2020 Sep;64(8):1210-1217. doi: 10.1111/aas.13599. Epub 2020 Apr 28. PMID 32270496